CLINICAL TRIAL: NCT04082845
Title: The Effect of Web-Based Training on the Anxiety and Early Recovery Outcomes of Thyroidectomy Patients: Randomized Controlled Study
Brief Title: Effect of Web-Based Training With Thyroidectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Bahar CANDAS ALTINBAS, Research Assistant, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Nurse_thyro01
Record Dates: First submitted 2019-08-30; First posted 2019-09-09 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Thyroidectomy; Education; General Surgery; Patient
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Parallel Assessment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will be educated via a website that was created by the researchers.
  Interventions: Other: Education
- Control Group (No Intervention): The control group will take rutin patient care.

INTERVENTIONS:
Other: Education — Web-based patient education
  Arms: Experimental Group

SUMMARY:
This study evaluates the effect of an internet website, created by the nurse for the purpose of internet-based training related to perioperative period, on the anxiety and postoperative recovery measures (length of hospitalization, first oral feeding time, first mobilization time, first defecation time, first gas release, pain, nausea, vomiting, re-admission) of thyroidectomy patients. For this, while the experimental group will educate via the internet, the control group will take rutin care.

DETAILED DESCRIPTION:
Today, due to changing guidelines, current approaches, and new paradigms, the approach to thyroid surgery has become more sensitive and selective. Besides, thyroid surgery has increased due to the increase in thyroid cancer and early detection of thyroid nodules. In a comprehensive study conducted by the Thyroid Cancer Association with 2398 patients in 35 countries, it is found that 92.6% of the patients did not receive psychological support, 84.1% did not receive institutional information, and 63.0% did not receive written information about the disease or treatment. Thyroidectomy patients are known to experience postoperative complications and symptoms such as hypocalcemia, hoarseness, dysphagia, drowsiness, or restricted neck/shoulder movement. Therefore, informing thyroidectomy patients about the surgical process will facilitate the management of the process. In addition to this, due to the increasing use of the internet with the developing technology, the behaviors of the patients searching for information from the internet are increasing day by day. It has been found that the rate of searching for health information from the internet is 68-72% in the world. Under this scope, this study will evaluate the effect of the web-based training on with thyroidectomy patients

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years and old,
* had planned surgery,
* speaks and understands Turkish,
* are literate,
* learned to have surgery at least one day before surgery,
* had first thyroidectomy,
* had total bilateral thyroidectomy,
* had internet connection at home or phone and
* had computer tablet or smartphone.

Exclusion Criteria:

* are mentally handicapped,
* are visual, hearing and speech impaired and
* had psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Concentration of patient anxiety | 9 days
  Self reported anxiety intensity during surgical process that includes on the day of surgery and one week after surgery. State-Trait Anxiety Inventory will be used to evaluate the anxiety. The higher the score is the more anxiety.
Rate of length of hospitalization | 2 days
  It means that how long did the patients stay at the hospital during surgery? This measure record via questionnaire as day. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.
Rate of first feeding time after surgery | 2 days
  It is described that how many hours after surgery did the patients eat first? This measure record via questionnaire as day. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.
Rate of first mobilization time after surgery | 2 days
  How many hours after surgery did the patients walk first? This measure record via questionnaire as day. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.
Rate of first defecation time after surgery | 2 days
  How many hours after surgery did the patients deface first? This measure record via questionnaire as day. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.
Rate of first gas release time after surgery | 2 days
  How many hours after surgery did the patients release gas first? This measure record via questionnaire as day. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups
Concentration of pain after surgery | 2 days
  It means that what is the severity of the pain that the patients had in 24 hours after surgery. It evaluated with Visual Analog Scale. The most common style used in pain measurement uses a horizontal line measuring exactly 10 cm. The patient is asked to make a mark on this line (from 0 to 10), then the line is measured and recorded in millimeters or centimeters. The higher the score is the more severe the pain. The severity of the pain compared between groups as average
Concentration of nausea after surgery | 2 days
  It is the severity of the nausea that the patients had in 24 hours after surgery. It evaluated with Visual Analog Scale. The patient is asked to make a mark on the line (from 0 to 10), then the line is measured and recorded in millimeters or centimeters. The higher the score is the more severe the nausea. The severity of the nausea compared between groups as average
Rate of vomiting after surgery until the discharge | 2 days
  It means that how many times did patients vomit until the discharge. It evaluated as number via questionnaire. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.
Number of Participants with re-admission after discharge | 9 days
  It shows that how many patients are re-admitted to the hospital in one week after discharge It evaluated as number via questionnaire. The minimum, maximum, median, 25th and 75th quartile were evaluated for each group and compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Candas Altınbas, PhD, Principal Investigator — Karadeniz Technical University
Locations (1):
- Bahar Candas Altinbas, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No